CLINICAL TRIAL: NCT06537700
Title: OnaBotulinumtoxin-A Effectiveness Evaluation in Chronic Migraine Patients with Short or Long Disease History: an Italian Multicentric Study (the BACH Study)
Brief Title: OnaBotulinumtoxin-A in Chronic Migraine Patients with Short or Long Disease History (the BACH Study)
Acronym: BACH
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Sponsor
Other Study IDs: 001.23(02.23) OSS; Fondazione PCBM (Other: Fondazione Policlinico Campus Bio-Medico)
Record Dates: First submitted 2024-07-17; First posted 2024-08-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Migraine
Keywords: Chronic migraine; OnabotulinumtoxinA; Migraine prevention; Disease duration; Psychiatric comorbidities
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group1 (>=10years) and Group1 (<10years): Patients will be divided into 2 groups according to their CM history (duration): A) those from 1 to 9 years and B) those with 10 or more years of CM history.
  Interventions: Drug: OnabotulinumtoxinA OBT-A

INTERVENTIONS:
Drug: OnabotulinumtoxinA OBT-A — Patients will be re-evaluated every 3 months, at each OBT-A cycle, during the whole year of treatment. Every evaluation patients will show their diary of headaches with monthly migraine and headache days and acute medications taken.

SUMMARY:
The goal of this observational prospective multicentric study, 12 months duration is to investigate whether the history of Chronic Migraine and, more precisely, its duration for over or less than 10 years, can predict OBT-A treatment effectiveness.

Since CM patients may have a complex psychopathological profile and psychiatric symptoms represent a bad prognostic factor influencing treatment effectiveness, the present study will also aim at evaluating if the psychopathological profile of the enrolled patients may influence the outcome.

DETAILED DESCRIPTION:
Onabotulinumtoxin-A (OBT-A) is a worldwide approved preventive treatment for patients suffering from Chronic Migraine (CM, 1.3, ICHD III 2018). Its effectiveness in reducing headache frequency and disability has been demonstrated by two well-designed phase III clinical trials, PREEMPT 1 and 2 and, more recently, by some real-life studies.

However, the use of OBT-A in the real world clinical practice has been still raising some issues: i.e. searching for more adequate patients' selection, when discontinuing the OBT-A treatment and when resuming it, finding associated patients' psychopathological profile possibly influencing the treatment, and so on. Moreover, finding some indicators of good or bad prognosis coming from OBT-A real-life experience could be of help for the clinicians to individuate the best candidates to the treatment.

The aim of the present study is mainly to investigate whether the history of Chronic Migraine and, more precisely, its duration for over or less than 10 years, can predict OBT-A treatment effectiveness. In other words, the study will aim to establish whether starting OBT-A treatment earlier in CM patients' life could make it more effective.

Since psychiatric symptoms may represent prognostic factors influencing treatment effectiveness, the present study will also aim at evaluating if the psychopathological profile of the enrolled patients may influence the outcome.

Consecutive CM patients treated in Italian tertiary level Headache Centers and classified according to CM history (shorter/longer than 10 years) will be enrolled.

Aims

To compare OBT-A treatment effectiveness in patients with shorter (1-9 yrs) and longer (10 or longer) years history of CM, in terms of:

* monthly migraine (MMD) or headache (MHD) days
* monthly acute medications (MAM)
* disability scales (Headache Impact Test, HIT-6; Migraine Disability Assessment MIDAS questionnaire) scores
* pain intensity and quality

Objectives

* to investigate whether the history of Chronic Migraine (over or less than 10 years) can predict OBT-A treatment effectiveness
* to find possible indicators of good or bad prognosis coming among psychiatric comorbidities of the enrolled patients

Consecutive CM patients (according to ICHD-3 1.3) treated in Italian headache centers, undergoing OBT-A, will be enrolled.

Methods All patients will fill a headache diary to report MMDs and acute medications taken every month.

Disability will be assessed by means of HIT-6 and MIDAS. Moreover, the intensity and quality of perceived pain will be evaluated by means of Numerical Rating Scale (NRS), 11-point Box Scale (BS-11), Present Pain Intensity (PPI), Behavioral Rating Scale (BRS-6) e Short-form McGill Pain Questionnaire (SF-MPQ).

The psychopathological profile will be evaluated at different times of the study by means of the following psychological questionnaires: Beck Depression Inventory (BDI-II), State-Trait Anxiety Inventory (STAI-Y), Toronto Alexithymia Scale (TAS-20).

At enrolment (T0), before starting the treatment, patients will have to fill a questionnaire about the previous 3 months (screening phase) including:

* MMD and MHD
* MAM
* NRS, BS-11, PPI, BRS-6 e SF-MPQ scales
* MIDAS e HIT-6 scale
* BDI-II, STAI-Y, TAS-20 questionnaires After completing the diary and scales above, patients will receive OBT-A treatment according to PREEMPT protocol.

Patients will be divided into 2 groups according to their CM history (duration): A) those from 1 to 9 years and B) those with 10 or more years of CM history.

Patients will be re-evaluated every 3 months, at each OBT-A cycle, during the whole year of treatment. At every evaluation time patients will show their diary of headaches with MMD and MAM taken.

At T3 and T9 (3 and 9 months respectively after T0), patients will fill the questionnaire including MMD and MAM taken in the previous 3 months, pain evaluation scales, MIDAS e HIT-6 scales.

At T6 and T12 (6 and 12 months respectively from T0, T12 being the final evaluation) patients will have to fill all questionnaires/scales as at T0.

Outcomes Primary endpoint Change in the mean number of MMD (or MHD) from baseline to months 6 through 12 between groups

Secondary

1. 50% or greater reduction in MMD from baseline to months 6 through 12 between groups
2. change in the number of MAM from baseline to months 6 through 12 between groups
3. change in pain intensity and quality scores from baseline to months 6 through 12 between groups
4. change in terms of psychological profile (STAI-Y, TAS-20 scales) in the stratified subgroups based on Z score of BDI-II scale (< 0 ≥ 1,8) between groups

Statistical analysis The data will be collected in an electronic database in anonymous form that will be protected by a password for each participant center.

On the basis of primary outcome (change during the follow-up vs. baseline of MMD), a general linear model with mixed effects will be applied, which will allow to evaluate, considering the within-subject dependencies and allowing to use all the observations available for each subject (even if for example the measurement of a subject at the time Tx should be missing), the interaction time X group and estimate if and when during follow-up a significant difference between the two groups will occur. According to a previous study (Vernieri et al, Headache 2019), the distribution of MMD is expected to follow a Gaussian distribution, therefore the general linear model will be a mixed-effects ANOVA. For some of the other variables (such as the number of analgesics or MIDAS) a generalized model will be applied to take into account the non-Gaussian nature of their distributions.

The sample size has been predefined according to the primary outcome with the following approach. Thanks to the previous study (Vernieri et al, 2019), it was possible to estimate the standard deviations (SD) of the changes of MMD between baselines and subsequent times. The maximum standard deviation was observed between baseline (T0) and T4 (1 year) and was 8 (with very similar values in two independent centers: 7.8 and 8.2). Since this SD was estimated on 100 patients, the 95% confidence interval for SD is 7.0-9.3. In order to avoid underestimation of the variability of the primary outcome, we have therefore set SD equal to the upper limit of the confidence interval built on the maximum SD found of the variations (vs. baseline) during the follow-up and that is SD=9.3.

In the following table it is reported the sample size required to have a power of 90% to recognize as statistically significant (at two-tails alpha level set at 0.05) the differences between the expected decreases specified in the first two columns. Since the evaluation times at follow-up will be 4 (T3, T6, T9, T12), the probability of error of type I has been divided by 4, in order to keep the overall alpha error below 5%.

In the cited study a decrease after 6 months of treatment (and confirmed at 12 months) of about 7 days of migraine/month was observed. This absolute decrease corresponded to a percentage change of about 30-35%. The hypothesis is that chronic patients from more than 10 years may benefit less from treatment and, in particular, that between the two groups there is a difference in efficacy of 4 (hypothesis 1) and 6 (hypothesis 2) days/month.

Hypothesis 1 Expected pre-post decrease Group1 (>=10y) 5 (SD=9.3) Expected pre-post decrease Group1 (<10y) 9 (SD=9.3) Power (1-b) 90% a (two-tails) 0.0125 N Group1 115 N Group1 115

Hypothesis 2 Expected pre-post decrease Group1 (>=10y) 4 (SD=9.3) Expected pre-post decrease Group1 (<10y) 10 (SD=9.3) Power (1-b) 90% a (two-tails) 0.0125 N Group1 52 N Group1 52

With these numbers it is also possible to calculate that there will be a probability of 90% to recognize as statistically significant (at alpha level 0.05) standardized effect size f=0.08 (hypothesis1) and f=0.12 (hypothesis 2) for the interaction Time X Group. The calculation for the interaction was based on an ANOVA with 4 repeated measurements after T0 (T3, T6, T9, T12), assuming the same correlation between the baseline follow-up assessments observed in the study by Vernieri et al, 2019 and applying a correction for lack of sphericity epsilon=0.9. Considering that f=0.10 is conventionally classifiable as "small", the indicated number of values therefore allow to be sensitive to small variations (even if clinically relevant).

Reference

Vernieri et al. Onabotulinumtoxin-A in Chronic Migraine: Should Timing and Definition of Non-Responder Status Be Revised? Suggestions From a Real-Life Italian Multicenter Experience. Headache. 2019 Sep;59(8):1300-1309.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years-old
* Chronic Migraine defined according to 1.3 ICHD-3
* Informed consent

Exclusion Criteria:

* secondary headache
* Onabotulinumtoxin-A in the previous 3 months
* pregnancy or breastfeeding
* detoxification protocol for Medication Overuse Headache in the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive CM patients (according to ICHD-3 1.3) treated in 8 Italian headache centers, undergoing OBT-A, will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Monthly Migraine Days (MMD), Monthly Headache Days (MHD) | baseline to months 6 through 12
  Change in the mean number of MMD (and MHD) from baseline to months 6 through 12 between groups

SECONDARY OUTCOMES:
50% or greater reduction in monthly migraine days (MMD) | from baseline to months 6 through 12 between groups
  50% or greater reduction in MMD (50% responder rate)
Number of monthly acute medications (MAM) | from baseline to months 6 through 12 between groups
  Change in the number of MAM
Pain intensity score, Numerical Rating Score NRS | from baseline to months 6 through 12 between groups
  Change in pain intensity score (11-point scale for self-report of pain, where 0 = no pain and 10 = extreme pain/worst possible pain.)
Pain intensity score, Present Pain Intensity PPI | from baseline to months 6 through 12 between groups
  Change in pain intensity score (recorded as a number from 1 to 5, in which each number is associated with the following words: 1 mild, 2 discomforting, 3 distressing, 4 horrible, 5 excruciating, i.e. higher figure means the worst outcome)
Pain quality score, the 6-point Behavioral Rating Scale (BRS-6) | from baseline to months 6 through 12 between groups
  The BRS-6 scale describes the limitations of activities because of pain and it is articulated in 6 grades: 1. No pain, 2. Pain is present but does not limit my activities, 3. Can do most activities, 4. Unable to do some activities, 5. Unable to do most activities, 6. Unable to do any activities
Pain quality score, the short-form McGill pain questionnaire SF-MPQ | from baseline to months 6 through 12 between groups
  The main component of the SF-MPQ consists of 15 pain quality descriptors (11 sensory = throbbing, shooting, stabbing, sharp, cramping, gnawing, hot-burning, aching, heavy, tender, splitting and 4 affective = tiring-exhausting, sickening, fearful and cruel-punishing) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe
Disability score, 6-item Headache Impact Test | from baseline to months 6 through 12 between groups
  Each of the six questions of the HIT-6 receives a score from 6-13. The final HIT-6 score can range from 36 to 78. A higher score indicates more disability due to headache
Disability score, Migraine Disability Assessment MIDAS questionnaire | from baseline to months 6 through 12 between groups
  The MIDAS score measures disability in migraine patients every 3 months, global score minimum 0, maximum 270, higher score means worse outcome; 4 grades of disability: 0 to 5 - MIDAS Grade I, Little or no disability 6 to 10 - MIDAS Grade II, Mild disability 11 to 20 - MIDAS Grade III, Moderate disability 21+ - MIDAS Grade IV, Severe disability
Psychological profile in terms of Trait subtest of State-Trait Anxiety Inventory (STAI) | from baseline to months 6 through 12 between groups
  Change of STAI-Y score (Spielberger et al., 1983), a 20 multiple-choice items self-report questionnaire for measuring anxiety disorder (each item from 1=lower, 4=higher anxiety level, i.e. global score minimum 20, maximum 80, higher score means worse outcome)
Psychological profile in terms of Beck Depression Inventory-II Edition, BDI-2 | from baseline to months 6 through 12 between groups
  Change of BDI-2 score (Beck et al., 1996), a 21 multiple-choice questions self-report inventory to measure the severity of depression (each item from 0=no symptoms, 3=higher level, the global score ranges from 0 to 63, where higher score means worse outcome)
Psychological profile in terms of Toronto Alexithymia Scale TAS-20 | from baseline to months 6 through 12 between groups
  Change of TAS-20 score (Bressi et al., 1996) a 20 multiple-choice items self-report inventory for evaluating difficulties to identify and describe emotions (Score 20-100, where 60 or higher indicates alexithymia)

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Università Politecnica delle Marche, Ancona
  - Università Studi dell'Aquila, L’Aquila
  - IRCCS Istituto Auxologico Italiano, Milan
  - Istituto Neurologico Besta, Milan
  - Fondazione Policlinico Campus Bio-Medico, Roma
  - Policlinico Tor Vergata, Roma

REFERENCES:
- [Background] Vernieri F, Paolucci M, Altamura C, Pasqualetti P, Mastrangelo V, Pierangeli G, Cevoli S, D'Amico D, Grazzi L. Onabotulinumtoxin-A in Chronic Migraine: Should Timing and Definition of Non-Responder Status Be Revised? Suggestions From a Real-Life Italian Multicenter Experience. Headache. 2019 Sep;59(8):1300-1309. doi: 10.1111/head.13617. Epub 2019 Aug 27. PMID 31454075
- See also: link to reference — https://pubmed.ncbi.nlm.nih.gov/31454075/